CLINICAL TRIAL: NCT01571791
Title: A Randomized Study of the Effects of Perioperative i.v. Ketorolac-lidocaine on the Hemodynamic Response in the Patients With Valvular Heart Diseases During Cesarean Delivery
Brief Title: Perioperative Ketorolac-lidocaine in the Patients With Valvular Heart Diseases During Cesarean Delivery
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: No enough recruited cases
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed R El Tahan, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R/41
Record Dates: First submitted 2012-03-31; First posted 2012-04-05 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Valve Heart Disease; Elective Cesarean Delivery
Keywords: Ketorolac; lidocaine; valvular hear diseases; cesarean section
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group SF (Placebo Comparator): either saline infusion and intravenous fentanyl boluses
  Interventions: Drug: Placebo
- group KL (Active Comparator): ketorolac-lidocaine infusion and intravenous saline boluses
  Interventions: Drug: Ketorolac-Lidocaine

INTERVENTIONS:
Drug: Placebo — to receive saline infusion and intravenous fentanyl boluses, at 30 min before induction of anesthesia
  Arms: group SF
Drug: Ketorolac-Lidocaine — receive ketorolac-lidocaine infusion and intravenous saline boluses , at 30 min before induction of anesthesia
  Arms: group KL

SUMMARY:
Rheumatic heart valve diseases are prevalent among the young people in Egypt secondary to the socioeconomic conditions. The goal of anesthetic management of these patients is maintenance of sinus rhythm, systemic blood pressure, preload, coronary perfusion, and cardiac output. Many women still prefer general anesthesia rather than regional techniques at the author's country.

The pharmacological modifications of the sympathetic response to tracheal intubation and surgical stimulation using opioids have adverse effects on the neonatal outcome after cesarean delivery. The authors have demonstrated in their previous studies the safety of both perioperative infusion of both of ketorolac and lidocaine in the attenuation of the hemodynamic and hormonal responses of tracheal intubation and surgery during cesarean delivery with favorable neonatal outcome and without added risk of perioperative bleeding. Therefore, the authors reported successful anesthetic management of a parturient with infective endocarditis on top of rheumatic mitral valve disease with use of paracetamol-lidocaine-ketorolac-propofol anesthesia.

The investigators hypothesize that the perioperative use of ketorolac-lidocaine would reduce the maternal hemodynamic responses to intubation and surgery without any harmful effects on mother or baby during uncomplicated cesarean delivery in the parturients with valvular hear diseases.

The investigators are aiming to compare the effects of ketorolac-lidocaine and fentanyl on surgical stress responses, intraoperative fentanyl and vasoactive drugs consumption and neonatal outcome during cesarean delivery in the parturients with valvular hear diseases.

DETAILED DESCRIPTION:
All parturients will receive oral ranitidine 150 mg on the night and the morning of surgery and 30 mL of 0.3 mol/L sodium citrate, 15 min before induction.

All operations will be performed by the same obstetricians. Voluven 6% solution 7 mL/kg will be infused over 30 min. Left uterine displacement will be maintained before induction. All routine medications except angiotensin-converting enzyme inhibitors will be continued until the morning of the operation.

All patients will be monitored with pulse oximetry, non-invasive blood pressure and five leads electrocardiography (leads II and V5). A radial artery catheter and a central venous catheter will be placed under local anesthesia before induction. On-screen pressure tracing will be used to determine end-expiration, and the CVP will be averaged over three respiratory cycles to eliminate respiratory artifacts. All staff in the operating room will be unaware of the randomization code.

After pre-oxygenation for 5 min, a rapid sequence induction will be performed with propofol 1-2.5 mg/kg and suxamethonium 1.5 mg/kg. Cricoid pressure will be applied, laryngoscopy will be performed after the 1-min blood pressure recording, and tracheal intubation will be completed before the 2-min reading. Anesthesia will be maintained with end-tidal concentrations of 2-2.5% of sevoflurane, in combination with 50% nitrous oxide in oxygen and cisatarcurium 0.1-0.2 mg/kg. The patients' lungs will be ventilated to maintain an EtCO2 of 4-4.6 kPa.

After the umbilical cord was clamped, infusion of 5-10 U oxytocin, midazolam 0.05 mg/kg and fentanyl 1-2 µg/kg will be given and nitrous oxide will be increased to 70%. Sevoflurane will be discontinued at the start of skin closure and the nitrous oxide will be discontinued after the last skin suture will be applied. At the end of surgery, residual neuromuscular block will be antagonized with neostigmine 50 µg/kg and atropine 20 µg/kg, and trachea will be extubated.

Intraoperative hypertension, defines as increase in mean arterial blood pressure (MAP) >= 25% of baseline for more than 1 min, with or without associated tachycardia (defined as HR value > 20% of the baseline value > 2 min) will be treated with IV boluses of fentanyl (1μg/kg). If blood pressure levels do not reach at least 20% of baseline levels after 5 min, slow intravenous administration of labetalol 20 mg will be considered. In the presence of hypotensive episodes (MAP decreased to <= 60 mmHg >= 2-3 min) and CVP < 8 mmHg, 5-7 ml/kg of 6% hydroxyethyl starch 130/0.4 will be given. In the presence of MAP ≤ 60 mmHg, and CVP > 10 mmHg, repeated bolus doses of ephedrine 5 mg will be given 5 min apart from each dose. Tachycardia ≥ 20% from the baseline values for ≥ 1 min will be treated with boluses of esmolol 20 mg.

ELIGIBILITY:
Inclusion Criteria:

* 90 ASA II & IV women
* with documented valvular heart disease
* uncomplicated
* singleton pregnancies of at least 36 weeks' gestation
* scheduled for elective cesarean delivery
* under general anesthesia

Exclusion Criteria:

* history of un-controlled hypertension
* ischemic heart disease
* left-ventricular ejection fraction less than 45%
* severe pulmonary hypertension
* critical aortic stenosis
* peripheral vascular disease
* thyrotoxicosis
* neurological diseases
* hepatic diseases w
* renal diseases
* allergy
* those requiring preoperative inotropic, vasopressor,
* mechanical circulatory or ventilatory support
* pregnancy-induced hypertension
* evidence of intrauterine growth restriction
* fetal compromise.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-06; Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
hemodynamics | Baseline, intraoperative, an expected average of 1 hour
  changes in blood pressures and heart rate

SECONDARY OUTCOMES:
changes in fentanyl consumption | intraoperative, an expected average of 1 hour
  Intraoperative fentanyl consumption
perioperative bleeding | intraoperative, an expected average of 1 hour, up to 24 hours after surgery
  Intra-operative blood loss will be assessed by measuring blood in the suction bottle minus the sonographically estimated amniotic fluid volume, visual estimate of blood on drapes and floor and weighing swabs after use. Postoperative transfusion requirements and blood loss will be estimated as previously reported by Huang et al. from inspection of the perineal pad (0: small; 1: moderate; 2: large). Haematocrit values will be recorded before and 48 h after surgery.
neonatal outcome | up to 24 hours after delivery
  Neonatal umbilical artery and umbilical vein blood pH, gas tensions, and base excess values.
  Apgar scores at 1 and 5 min, and newborns' blood pressure, heart rate, temperature, arterial oxygen saturation, and the Neurologic and Adaptive Capacity Score (NACS) will be recorded at 15 min, 2 and 24 h after delivery.
uterine tone | intraoperative, an expected average of 1 hour
  The obstetrician will assess uterine tone by palpation every 5 minutes after delivery of the placenta using a 10-cm VAS (0: well contracted; 10: completely relaxed). If uterine tone remains unsatisfactory after 3 min, an additional 5 U bolus of oxytocin will be administered.
postoperative pain | up to 24 after surgery
  a 10-cm VAS at rest and on movement (0: no pain; 10: worst pain imaginable) 0, 1, 2, 4, 6, 8, 10 and 12 h after surgery. For postoperative pain relief intravenous 100 mg will be given when VAS scores are 5 or more at rest, or 7 or more on movement, or if the patient requests additional analgesia. The time to first request for analgesia and the number of subjects receiving tramadol during the first 12 h will be recorded.
perioperative side effects | up to 24 after surgery
  perioperative side effects includes arrhythmia, sedation, nausea and vomiting, light-headedness, headache, perioral numbness, tunnel vision, or seizures

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospitals, Al Mansurah, DK, Egypt